CLINICAL TRIAL: NCT05332756
Title: Long-term Outcomes of Conservative Management in Patients with Moyamoya Disease and Their First-degree Relatives
Brief Title: Long-term Outcomes of Conservative Management in Patients with Moyamoya Disease and Their First-degree Relatives (LAMORA)
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2021-186-02
Record Dates: First submitted 2022-03-31; First posted 2022-04-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya Disease; Conservative management; Long-term follow-up; First-degree relatives
MeSH Terms: conditions — Moyamoya Disease | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Moyamoya disease patients
  Interventions: Other: Conservative management
- First-degree relatives of patients with Moyamoya Disease

INTERVENTIONS:
Other: Conservative management — Patients and their first-degree relatives will be medically treated with antiplatelets, antiepileptics, antihypertensives and vasodilators depending on the presentation.
  Groups: Moyamoya disease patients

SUMMARY:
The purpose of this study is to investigate the long-term outcomes of conservative management in patients with moyamoya disease and their first-degree relatives, and provide potential pathogenesis of moyamoya disease.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a chronic occlusive-stenosis cerebrovascular disease that characterized by the stenosis of internal carotid artery termination and the formation of net-like vessel. It is a multifactorial disease caused by genetic, inflammatory, immunological and other environmental factors. The specific pathogenesis of MMD is still unclear. The treatment modalities of revascularization and conservative management have been used in patients with MMD. However, the long-term outcomes of MMD with conservative management remain unknown. Also, some first-degree relatives who are carriers of genetic variants occasionally manifest with intracranial arterial stenosis. Therefore, it is significant to detect the long-term outcomes of conservative treatment in MMD patients and their first-degree relatives, and thus provide potential pathogenesis of MMD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 2-60 years;
2. A clinical diagnosis of moyamoya disease, including unilateral and bilateral disease.
3. Patients are medically treated with antiplatelets, antiepileptics, antihypertensives and vasodilators depending on the presentation.
4. Capable of understanding the purpose and risk of the study and has signed the informed consent. If the participant is not capable of this at the time of enrollment, a legally authorized representative will provide written informed consent in accordance with all regulations.
5. Ability to comply with study follow-up.

Exclusion Criteria:

1. Concomitant other diseases, including systemic vasculitis, neurofibroma, meningitis, sickle cell disease, down's syndrome, and previous basilar radiotherapy.
2. Patients with cardiogenic embolism, including a history of atrial fibrillation, valvular disease or cardiac valve replacement.
3. Patients are allergic to the contrast agents.
4. Patients are treated with direct, indirect, or combined revascularization depending on the presentation.
5. Physical or subjective failure to cooperate with the examination or serious comorbid diseases.
6. Patients are unable or unlikely to return for follow-up visits.
7. Any other reasons that, in the opinion of the investigators, make the participant unsuitable for enrollment.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Consecutive patients diagnosed with MMD in Beijing Tiantan Hospital will be recruited. Eligibility will be determined through a checklist of inclusion and exclusion criteria. Relatives will be recruited from the first-degree relatives of patients with MMD.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular events | 6 months
Cerebrovascular events | 1 year
Cerebrovascular events | 2 years
Cerebrovascular events | 5 years

SECONDARY OUTCOMES:
Identification of RNF213 variants | Baseline
Unfavorable neurological outcome (mRS>2) | 6 months, 1 year, 2 years, and 5 years during follow-up
Change in cerebral perfusion status as assessed by CTP | Baseline, 6 months, 1 year, 2 years, and 5 years during follow-up
Change in immunological, inflammatory, angiogenesis biomarkers of peripheral blood | Baseline, 1 year, 2 years, and 5 years during follow-up
  Serum, plasma, RNA, immune cells and cytokines
Change in angiographic features as assessed by CTA | Baseline, 6 months, 1 year, 2 years, and 5 years during follow-up
Change in angiographic characteristics as assessed by MRA | Baseline, 1 year, 2 years, and 5 years during follow-up
Change in radiological characteristics as assessed by HR-MRI | Baseline, 1 year, 2 years, and 5 years during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No